A Randomized, Double-Blind, Vehicle-Controlled Study to evaluate the Efficacy and Safety of Topical Administration of FMX101 for 12 Weeks in the Treatment of Moderate-to-Severe Acne Vulgaris (Study FX2017-22)

Protocol Synopsis

NCT03271021

Date: 22 June 2017



## **Synopsis**

| Name of Sponsor/Company: Foamix Pharmaceuticals, Inc. | Individual Study Table Referring to Part of the Dossier: | (For National Authority<br>Use Only) |
|---|---|---|
| Name of Finished Product:<br>FMX101 | Volume: | |
| Name of Active Ingredient: | Page: | |
| Minocycline hydrochloride | | |
| Title of Study: | A Randomized, Double-Blind, Vehicle-Controlled Study to Evaluate the Efficacy and Safety of Topical Administration of FMX101 for 12 Weeks in the Treatment of Moderate-to-Severe Acne Vulgaris (Study FX2017-22) | |
| Protocol No: | FX2017-22 | |
| Study Centers: | Multicenter (approximately 80 sites in the USA) | |
| Publication (reference): | None | |
| Phase of Development: | 3 | |
| Objectives: | <ul> <li>To evaluate the efficacy in the treatment of acne compared to vehicle of topical FMX101 4% administered daily for 12 weeks.</li> <li>To evaluate the safety compared to vehicle of topical FMX101 4% administered daily for 12 weeks.</li> </ul> | |
| Study Design and Methods: | This is a randomized, multicenter, double-blind, vehicle-controlled, 2-arm study to evaluate the safety and efficacy over 12 weeks of FMX101 topical foam containing 4% minocycline compared to vehicle in the treatment of subjects with moderate-to-severe facial acne vulgaris. Qualified subjects will be randomized, stratified by investigational site, in a 1:1 ratio (active:vehicle) to receive 1 of the following 2 treatments: | |
| | FMX101 4% minocycline foam | |
| | Vehicle foam | |
| | Subjects will apply (or have it applied) the assigned study drug topically once daily for 12 weeks as directed. Subjects will be advised to apply the study drug at approximately the same time each day, preferably about 1 hour before bedtime. Both the Investigator and subject will be blinded to the study drug identity. | |
| | Subjects will return for visits at Weeks discretion of the clinic staff, for the constaff, visits can be scheduled to occur anominal scheduled date for the Weeks before or after for the Weeks 9 and 12 (acne lesion counts and Investigator G performed at Screening/Baseline and a | nvenience of subjects or clinic<br>3 days before or after the<br>1, 3, and 6 visits and 7 days<br>visits. Efficacy evaluations<br>lobal Assessment [IGA]) will be |



| Number of Subjects (planned): | The planned enrollment is approximately 1500 subjects. |
|---|---|
| Diagnosis and Main<br>Criteria for Inclusion: | Healthy male or non-pregnant females, aged ≥9 years, with a clinical diagnosis of moderate-to-severe facial acne vulgaris characterized by (subjects are permitted to also have acne on other parts of the body): • 20 to 50 inflammatory lesions (papules, pustules, and nodules) • 25 to 100 non-inflammatory lesions (open and closed comedones) • No more than 2 nodules on the face • An IGA score of moderate (3) to severe (4) |
| Test Product, Dose and<br>Mode of Administration: | FMX101 minocycline foam 4%. Topical application, once daily to the face, for 12 weeks. |
| Reference Therapy: | Vehicle foam. Topical application, once daily to the face, for 12 weeks. |
| Study Duration: | Subject participation in the study will be up to 18 weeks: up to 6 weeks for Screening and Baseline, and 12 weeks of study treatment. |
| Endpoints and Outcomes: | Efficacy Evaluations The efficacy assessments will include lesion counts and the IGA at Baseline and at Weeks 3, 6, 9, and 12. |
| | Safety Evaluations The safety assessments will include adverse events (volunteered, observed, and elicited by general questioning in a non-suggestive manner), physical examinations, vital signs, local skin assessment scores (including erythema, dryness, peeling, and hyperpigmentation), and clinical laboratory test results. |
| Statistical Methods: | |